CLINICAL TRIAL: NCT00230386
Title: The Role of MRI Perfusion to Detect Locally Recurrent or Persistent Disease in Prostate Carcinoma Treated With Radiation Therapy - A Pilot Study
Brief Title: Role of Magnetic Resonance Imaging (MRI) Perfusion to Detect Disease in Prostate Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 03-0272-CE
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2005-09

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Device: MRI

SUMMARY:
This is a pilot study of 50 patients to establish whether there is a potential role for MRI perfusion in the detection of locally recurrent or persistent prostate carcinoma after previous treatment with radiotherapy. All subjects will be patients who have had localised prostate cancer treated with radiotherapy and have already agreed to undergo a biopsy of the prostate to look at local control within the prostate as part of their management. The objective of the study is to establish whether there is a relationship between recurrent or persistent disease within the prostate and increased perfusion on MRI at these sites.

ELIGIBILITY:
Inclusion Criteria:

* Previously have had radical radiotherapy for localised prostate cancer
* Due to undergo routine post-treatment prostatic biopsies
* Suitable for MRI scan
* Adequate renal function
* No previous reaction to gadolinium
* Able to give informed consent
* No recent prostate biopsy within 6 weeks of enrolment
* Performance status (Eastern Cooperative Oncology Group [ECOG]) 0 or 1

Exclusion Criteria:

* Not suitable for MRI scan
* Previous reaction to gadolinium
* Impaired renal function
* Inability to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-05

PRIMARY OUTCOMES:
To determine whether there may be a role for MRI perfusion in the detection of recurrent or persistent prostatic cancer after previous radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network Princess Margaret Hospital, Toronto, Ontario, Canada